CLINICAL TRIAL: NCT01981486
Title: A Phase I, Placebo Controlled, Randomized, Subject-And Investigator-Blind, Sponsor-Open, Multiple Ascending Dose Study To Evaluate The Safety, Tolerability, And Pharmacokinetics Of PF-05180999 In Healthy Adult Volunteers
Brief Title: A Study Of The Safety, Tolerability, And Pharmacokinetics Of Multiple Doses Of PF-05180999 In Healthy Adults
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B3441008
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Migraine
Keywords: PF-05180999; safety; tolerability; pharmacokinetics; migraine; PDE2; cAMP; cGMP; cantharidin; blister; CYP3A induction
MeSH Terms: conditions — Migraine Disorders; Blister

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Drug: Placebo Tablets
- PF-05180999 (Experimental): Modified-release tablets of PF-05180999
  Interventions: Drug: PF-05180999 Tablets

INTERVENTIONS:
Drug: Placebo Tablets — BID modified-release tablets
  Arms: Placebo
Drug: PF-05180999 Tablets — BID modified-release tablets (20 to 240 mg BID)
  Arms: PF-05180999

SUMMARY:
PF-05180999 is a novel phosphodiesterase-2 (PDE2) inhibitor. The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of multiple doses of PF-05180999 administered twice daily over 14 days. Exploratory measures of PDE2 inhibition will also be evaluated in blood and blister fluid.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female (of non-childbearing potential) subjects between the ages of 18 and 55 years
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs)

Exclusion Criteria:

* Subjects with Gilbert's disease or screening laboratory test results that deviate from the upper and/or lower limits of the reference or acceptable range. The exception is that all liver function tests must not exceed the upper limit of normal.
* Subjects with evidence of, or history of, hepatic disorder, including acute or chronic hepatitis B or hepatitis C.
* Subjects with very light skin or very dark skin (at the discretion of the investigator).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 0-12 hours post-dose on Day 1
  Single dose Cmax
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0-12 hours post-dose on Day 1
  Single dose Tmax
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) | 0-12 hours post-dose on Day 1
  Single dose AUCtau
Maximum Observed Plasma Concentration at Steady-State (Cmax,ss) | 0-12 hours post-dose on Day 14
  Steady-state Cmax
Time to Reach Maximum Observed Plasma Concentration at Steady-State (Tmax,ss) | 0-12 hours post-dose on Day 14
  Steady-state Tmax
Minimum Observed Plasma Trough Concentration at Steady-State (Cmin,ss) | 0-12 hours post-dose on Day 14
  Steady-state Cmin
Area Under the Curve from Time Zero to End of Dosing Interval at Steady-State (AUCtau,ss) | 0-12 hours post-dose on Day 14
  Steady-state AUCtau
Apparent Oral Clearance (CL/F) | 0-48 hours post-final dose on Day 14
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) | 0-48 hours post-final dose on Day 14
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Plasma Decay Half-Life (t1/2) | 0-48 hours post-final dose on Day 14
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Accumulation Ratio (Racc) | 0-12 hours post-dose on Days 1 and 14
  Ratio of Day 14 AUCtau to Day 1 AUCtau
Amount Excreted in Urine (Ae) | 0-12 hours post-dose on Day 14
  Amount of drug excreted in urine
Percent of Dose Excreted in Urine (Ae%) | 0-12 hours post-dose on Day 14
  Percent of total dose excreted in urine
Renal Clearance (CLr) | 0-48 hours post-dose on Day 14
  Renal clearance is a quantitative measure of the rate at which a drug substance is removed from the blood via the renal route.

SECONDARY OUTCOMES:
Identification of metabolites of PF-05180999 in urine and plasma | 0-12 hours post-dose on Day 14
  Metabolite identification
Change from Baseline in Total Leukocyte Levels and Leukocyte Subpopulations in Blister Fluid and Blood | Day 13 and Day 14
  Leukocyte levels in blister fluid and blood
Change from Baseline in Cytokine Levels in Blister Fluid | Day 13 and Day 14
  Cytokine levels in blister fluid
Time-Averaged Area Under the Effect Curve (AUEC/t) for Platelet cGMP and cAMP | 0-12 hours post-dose on Day 1 and Day 14
  Time-averaged area under the effect curve
AUEC/t Ratio | 0-12 hours post-dose on Day 1 and Day 14
  Ratio of Day 14 AUEC/t to Day 1 AUEC/t
Urinary 6beta-hydroxycortisol/cortisol ratio | Day 14
  Urinary marker of CYP3A induction
Plasma 4beta-hydroxycholesterol/cholesterol ratio | Day 14
  Plasma marker of CYP3A induction

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3441008&StudyName=A%20Study%20Of%20The%20Safety%2C%20Tolerability%2C%20And%20Pharmacokinetics%20Of%20Multiple%20Doses%20Of%20PF-05180999%20In%20Healthy%20Adults